CLINICAL TRIAL: NCT07043686
Title: Effect of Cerebrolysin on Early Rehabilitation After Ischemic Stroke at the Department of Vascular Neurology and Intensive Neurological Therapy (KOVNINT), University Medical Centre Ljubljana
Brief Title: Cerebrolysin in Early Stroke Rehabilitation - Tertiary Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Matija Zupan, neurologist, MD, PhD, University Medical Centre Ljubljana
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CER-KOVNINT-2025
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Ischemic Stroke, Acute; Rehabilitation Outcome; Cerebrolysin
Keywords: Cerebrolysin; Acute Ischemic Stroke; Neuroplasticity; Neurorehabilitation; Action Research Arm Test; Slovenia
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Cerebrolysin Group (Experimental): The patients in Arm 1 will be treated with cerebrolysin and standard treatment.
  Interventions: Drug: Cerebrolysin treatment; Other: Standard treatment (including neurorehabilitation) of acute ischemic stroke
- Arm 2: Standard treatment only Group (Other): The patients in Arm 2 will receive standard treatment only.
  Interventions: Other: Standard treatment (including neurorehabilitation) of acute ischemic stroke

INTERVENTIONS:
Drug: Cerebrolysin treatment — The patients will receive Cerebrolysin treatment, 10 days consecutively, 30 ml/day, intravenous infusion diluted up to 100 ml of 0.9% saline in 15 minutes.
  Arms: Arm 1: Cerebrolysin Group
Other: Standard treatment (including neurorehabilitation) of acute ischemic stroke — "Standard treatment" entails acute ischemic stroke reperfusion treatment according to international guidelines and local policies, instituting secondary preventive treatment, a proper management of stroke risk factors and neurorehabilitation according to patient's needs: locomotor physiotherapy, occupation therapy, speech therapy, and neuropsychological assessment.

SUMMARY:
The study evaluates the effect and safety of Cerebrolysin administered during early rehabilitation in patients with moderate neurological impairment after acute ischemic stroke, conducted at the Department of Vascular Neurology and Intensive Neurological Therapy, UMC Ljubljana.

DETAILED DESCRIPTION:
Cerebrolysin is a neuropeptide preparation from porcine brain in an aqueous solution. The composition of 1 ml of the solution contains 215.2 mg of a low molecular weight fraction of polypeptides extracted from porcine brain (Cerebrolysin concentrate), which corresponds to at least 5.8 mg of peptide nitrogen (15%) and free amino acids (85%).

Cerebrolysin has been registered for many years for the treatment of cerebrovascular and neurodegenerative diseases, as well as traumatic brain injuries worldwide. Since the first approval, the treatment of ischemic stroke (IS) has progressed and new treatment concepts have been developed. In addition, the treatment of IS with Cerebrolysin has developed with different time windows, doses and duration of treatment. The main objective of this study is to determine the effectiveness of Cerebrolysin in early rehabilitation as an adjunct to standard treatment in a group of patients with moderate to severe neurological impairment after acute IS in specific KOVNINT conditions.

All patients will receive acute IS care according to local standards of care, which will not be changed or influenced by the study in any way. To assess the safety and efficacy of Cerebrolysin in practice at KOVNINT, the outcome of patients treated with Cerebrolysin will be compared to patients in the control group who will not receive Cerebrolysin.

The reason for conducting the study is to determine the effectiveness of Cerebrolysin treatment in patients with moderate to severe neurological deficits after acute IS at KOVNINT and to assess the impact of these parameters on the outcome of treatment, especially the effect on neurological impairment at discharge and 90 days after IS.

The aim of this study is to observe the safety and efficacy of Cerebrolysin in patients with moderate to severe neurological impairment after acute IS in the specific KOVNINT conditions. We will conduct an analysis of the use of Cerebrolysin as an adjunct to standard treatment and evaluate its efficacy in the early phase of IS, defined by neurological impairment at discharge and 90 days after IS.

Consecutive patients will be enrolled in the study over a specified period, with the investigator independently deciding to treat with Cerebrolysin within 7 days after IS after obtaining informed consent. Patients will be included whose clinical diagnosis of acute IS will be confirmed by imaging, with patients having moderate to severe neurological impairment, defined by an initial NIHSS score of 6-12. All patients will receive standard care for IS according to local treatment. Treatment standards will not be changed and they will not be affected by the study.

Cerebrolysin group: (15 patients) Patients who will be treated with Cerebrolysin will receive the drug according to the SmPC. Dosage 30 ml/day, 10 days. Administration by intravenous infusion (IV infusion). Administration procedure: The drug is diluted to a volume of 100 ml with 0.9% saline. The infusion time will be 15 min.

Patients will receive the drug in accordance with the regulations on sterility of the application. To ensure sterility, single-use infusion sets and cannulas are always used. The infusion is started as soon as possible after dilution.

Control group: (15 patients) Patients receiving all standard care for ICU and not receiving Cerebrolysin.

ELIGIBILITY:
Inclusion Criteria:

Being able to perform ARAT test Signed informed consent

Both sexes, age not specified

Acute ischemic stroke confirmed by imaging

NIHSS score 6-12

No prior stroke or disability (mRS 0 before stroke)

-

Exclusion Criteria:

Not being able to perform ARAT test

* Previous stroke or disability (mRS > 0)
* The patient unable to understand instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2027-07-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
90-day Action Research Arm Test (ARAT) Score change | 90 days post-stroke
  A standardized test after stroke to measure the function of the upper limb. Range of scores: 0-57, with higher scores meaning a better outcome.

SECONDARY OUTCOMES:
National Institute of Health Stroke Scale (NIHSS) at discharge and 90 days | 90 days
  NIHSS is standardized in stroke medicine for measuring neurological deficits after stroke; range of scores 0-42, higher scores mean a worse outcome
Modified Rankin Score (mRS) at day 90 | 90 days
  mRS is a functional global scale measuring the functional disability after stroke, widely accepted in international registries and trials of stroke, range 0-6, with higher scores meaning worse outcome
Extended Barthel index (EBI) 90 days post-stroke | 90 days
  EBI measures neurological improvement after stroke in activities of daily living, range 0-100, with higher scores meaning better outcome
The De Morton Mobility Index (DEMMI) Score 90 days | 90 days
  Mobility assessment in elderly population, range 0-100, with higher scores meaning a better outcome
Montreal Cognitive Assessment (MoCA) 90 days | 90 days
  MoCA is a screening tool for mild cognitive impairment, range 0-30, with higher scores meaning a better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Matija Zupan, MD, PhD, Principal Investigator — University Medical Centre Ljubljana
Locations (1):
- UMC Ljubljana - Department of Vascular Neurology and Intensive Neurological Therapy (KOVNINT), Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
De-identified clinical outcomes data for academic purposes

REFERENCES:
- [Background] van den Brule FA, Castronovo V, Menard S, Giavazzi R, Marzola M, Belotti D, Taraboletti G. Expression of the 67 kD laminin receptor in human ovarian carcinomas as defined by a monoclonal antibody, MLuC5. Eur J Cancer. 1996 Aug;32A(9):1598-602. doi: 10.1016/0959-8049(96)00119-0. PMID 8911124